CLINICAL TRIAL: NCT06127888
Title: Implementació de Recomanacions d'Exercici Per al Tractament de Les Cefalees primàries: Una aproximació Qualitativa a Les Unitats de Cefalea a Catalunya
Brief Title: Impementation of the Exercise Recommendations for the Treatment of Primary Headaches: A Qualitative Approach to the Headache Units in Catalonia
Acronym: RECEPTA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Fundació Universitària del Bages (Other)
Responsible Party: Sponsor
Other Study IDs: I-RECEPTA JPA003
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-11

CONDITIONS: Migraine; Headache; Chronic Headache
Keywords: Exercise therapy; Neurology; Headache units; Primary headaches; Physiotherapy
MeSH Terms: conditions — Migraine Disorders; Headache; Headache Disorders | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Unit of headache and neurological pain of the Hospital Vall d'Hebron (VHIR) - Barcelona: Neurologists, nurses, pharmacists, health managers, physiotherapists, and other healthcare professionals related to the headache unit.
  Interventions: Other: Interviews; Other: Surveys
- Unit of headaches and neuralgias of the Hospital de Sant Pau - Barcelona: Neurologists, nurses, pharmacists, health managers, physiotherapists, and other healthcare professionals related to the headache unit.
  Interventions: Other: Interviews; Other: Surveys
- Unit of headache of the Hospital Sant Joan de Déu - Althaia - Manresa: Neurologists, nurses, pharmacists, health managers, physiotherapists, and other healthcare professionals related to the headache unit.
  Interventions: Other: Interviews; Other: Surveys
- Unit of headache of the Hospital Universitari Arnau de Vilanova - Lleida: Neurologists, nurses, pharmacists, health managers, physiotherapists, and other healthcare professionals related to the headache unit.
  Interventions: Other: Interviews; Other: Surveys
- Group of work on headaches of the Hospital Clínic de Barcelona: Neurologists, nurses, pharmacists, health managers, physiotherapists, and other healthcare professionals related to the headache unit.
  Interventions: Other: Interviews; Other: Surveys
- Headache Unit of Hospital de Bellvitge - Barcelona: Neurologists, nurses, pharmacists, health managers, physiotherapists, and other healthcare professionals related to the headache unit.
  Interventions: Other: Interviews; Other: Surveys
- Headache Unit of Hospital del Mar - Barcelona: Neurologists, nurses, pharmacists, health managers, physiotherapists, and other healthcare professionals related to the headache unit.
  Interventions: Other: Interviews; Other: Surveys
- Headache Unit of Hospital de Germans Tries i Pujol - Can Ruti - Badalona: Neurologists, nurses, pharmacists, health managers, physiotherapists, and other healthcare professionals related to the headache unit.
  Interventions: Other: Interviews; Other: Surveys
- Headache Unit of Hospital Josep Trueta - Girona: Neurologists, nurses, pharmacists, health managers, physiotherapists, and other healthcare professionals related to the headache unit.
  Interventions: Other: Interviews; Other: Surveys

INTERVENTIONS:
Other: Interviews — Semi-structured interviews
Other: Surveys — Estructured survey

SUMMARY:
Therapeutic exercise, including aerobic activity and strength training, has shown promise in treating primary headaches with a moderate effect size, despite limited evidence. Implementation requires specialized professionals, infrastructure, and defined care pathways. These strategies are cost-effective for similar chronic pain conditions. More research is needed to better understand the varying effects on headache frequency, duration, and intensity in larger patient samples.

DETAILED DESCRIPTION:
Therapeutic exercise strategies (TES) includes modalities such as aerobic activity and strength training, which have been investigated as treatments for primary headache in recent years. These modalities have been previously summarized, and despite the fact that the body of evidence available is less than in other therapeutic modalities, this is increasing, and they are positioned as strategies with a moderate effect size and recommendation.

However, its implementation is not simple and requires resources, such as professionals with specialized training, infrastructure, and clearly defined care circuits. Conversely, these strategies have demonstrated cost-effectiveness in other chronic pain conditions with similar treatment and care demands.

It is of interest to increase knowledge in this area given that the size of the effect of these interventions is large, although it varies according to the analyzed variable and type of exercise modality. The reduction in days per month with headache or migraine, reduction in headache hours per month, or decrease in headache intensity has been demonstrated in a non-negligible number of patients, but larger samples are needed.

The present study aimed to determine the status of exercise recommendations in the headache units of the Catalan territory and to evaluate the possible fit of specialized physiotherapy for the treatment of patients with headaches within these units based on the opinion of the responsible members of these units and available resources.

Contact with the headache units of the Catalan territory will be made by email or telephone during November 2023.

Semi-structured interviews and a survey developed from the interviews with the members of the units will be conducted to determine the status of exercise recommendations in the headache units of the Catalan territory and to evaluate the possible viability of specialized physiotherapy for the treatment of patients with headaches.

A total of 8-12 interviews and 20-30 responses to the surveys were expected. These will include neurologists, nurses, pharmacists, managers, rehabilitation doctors, and physiotherapists linked to neurology services.

ELIGIBILITY:
Inclusion Criteria:

* Be part of the headache unit
* Be a part of a service related to the headache unit
* Be a healthcare practitioner, researcher, health manager or rehabilitation service manager.

Exclusion Criteria:

* Decline participation
* Unable to understand Catalan, Spanish or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neurologists, nurses, pharmacists, researchers, physical therapists, rehabilitation doctors, health manager of the headache unit or rehabilitation service connected to the headache unit.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Status of exercise prescription in primary headaches | During observation period from November 2023 to January 2024.
  Likert Scale from 1-5: (1) Not recommended, (2) occasionally recommended, (3) usually recommended, (4) occasionally recommended and supervised by a qualified professional, (5) usually recommended and supervised by a qualified professional. Through survey and interviews.
Viability of the exercise prescription in the headache units | During observation period from November 2023 to January 2024.
  List of necessary resources for implementing exercise for primary headache patients reported by headache units. Qualitative information from surveys and interviews.
Relevance of exercise as a strategy for the treatment of patients with primary headaches. | During observation period from November 2023 to January 2024.
  Likert 1-5: (1) Not interesting for headache management, (2) Low interest for headache management (3) Moderate interest for headache management (4) High interest for headache management (5) Absolute interest for headache management. Through survey and interviews.

SECONDARY OUTCOMES:
Create a survey for assessing headache unit resources. | During November 2023
  List of essencial items to be included in the headache unit survey. Discussed by consensus among authors.
Necessary material resources | During observation period from November 2023 to January 2024.
  List of material resources needed for implementing physiotherapy in the headache units. Identified through semi-structured interviews.
Necessary technological resources | During observation period from November 2023 to January 2024.
  List of technological resources needed for implementing physiotherapy in the headache units. Identified through semi-structured interviews.
Necessary human resources | During observation period from November 2023 to January 2024.
  List of human resources needed for implementing physiotherapy in the headache units. Identified through semi-structured interviews.
Necessary service resources | During observation period from November 2023 to January 2024.
  List of service resources needed for implementing physiotherapy in the headache units. Identified through semi-structured interviews.
Necessary additional resources | During observation period from November 2023 to January 2024.
  List of additional resources needed for implementing physiotherapy in the headache units. Identified through semi-structured interviews.
Acceptance to implementation therapeutic exercice strategies | December 2023
  Number of headache units that accepts to participate in a protocol to implement any of the therapeutic exercice strategies.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manresa, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Should be discussed with the participants

REFERENCES:
- [Result] Hanssen H, Minghetti A, Magon S, Rossmeissl A, Rasenack M, Papadopoulou A, Klenk C, Faude O, Zahner L, Sprenger T, Donath L. Effects of different endurance exercise modalities on migraine days and cerebrovascular health in episodic migraineurs: A randomized controlled trial. Scand J Med Sci Sports. 2018 Mar;28(3):1103-1112. doi: 10.1111/sms.13023. Epub 2018 Jan 8. PMID 29161767
- [Result] Kroll LS, Hammarlund CS, Linde M, Gard G, Jensen RH. The effects of aerobic exercise for persons with migraine and co-existing tension-type headache and neck pain. A randomized, controlled, clinical trial. Cephalalgia. 2018 Oct;38(12):1805-1816. doi: 10.1177/0333102417752119. Epub 2018 Jan 15. PMID 29333870
- [Result] Madsen BK, Sogaard K, Andersen LL, Tornoe B, Jensen RH. Efficacy of strength training on tension-type headache: A randomised controlled study. Cephalalgia. 2018 May;38(6):1071-1080. doi: 10.1177/0333102417722521. Epub 2017 Jul 27. PMID 28750588
- [Result] van Ettekoven H, Lucas C. Efficacy of physiotherapy including a craniocervical training programme for tension-type headache; a randomized clinical trial. Cephalalgia. 2006 Aug;26(8):983-91. doi: 10.1111/j.1468-2982.2006.01163.x. PMID 16886935
- [Result] Alvarez-Melcon AC, Valero-Alcaide R, Atin-Arratibel MA, Melcon-Alvarez A, Beneit-Montesinos JV. Effects of physical therapy and relaxation techniques on the parameters of pain in university students with tension-type headache: A randomised controlled clinical trial. Neurologia (Engl Ed). 2018 May;33(4):233-243. doi: 10.1016/j.nrl.2016.06.008. Epub 2016 Aug 1. English, Spanish. PMID 27491303
- [Result] Reina-Varona A, Madronero-Miguel B, Gaul C, Hall T, Oliveira AB, Bond DS, Fernandez-de Las Penas C, Florencio LL, Carvalho GF, Luedtke K, Varkey E, Kroll LS, Bevilaqua-Grossi D, Kisan R, La Touche R, Paris-Alemany A. Therapeutic Exercise Parameters, Considerations, and Recommendations for Migraine Treatment: An International Delphi Study. Phys Ther. 2023 Oct 3;103(10):pzad080. doi: 10.1093/ptj/pzad080. PMID 37410390
- [Result] Miyamoto GC, Lin CC, Cabral CMN, van Dongen JM, van Tulder MW. Cost-effectiveness of exercise therapy in the treatment of non-specific neck pain and low back pain: a systematic review with meta-analysis. Br J Sports Med. 2019 Feb;53(3):172-181. doi: 10.1136/bjsports-2017-098765. Epub 2018 Apr 20. PMID 29678893
- [Result] Del Llano Senaris JE, Correia NN, Logusso LG, Errea Rodriguez M, Bringas Roldan C. [The indirect costs of tension type headache. A systematic literature review]. Aten Primaria. 2022 Mar;54(3):102238. doi: 10.1016/j.aprim.2021.102238. Epub 2022 Jan 22. Spanish. PMID 35077913
- [Result] Salazar A, Berrocal L, Failde I. Prevalence of Migraine in General Spanish Population; Factors Related and Use of Health Resources. Int J Environ Res Public Health. 2021 Oct 23;18(21):11145. doi: 10.3390/ijerph182111145. PMID 34769668
- [Result] Jimenez-Trujillo I, Lopez-de-Andres A, Del Barrio JL, Hernandez-Barrera V, Valero-de-Bernabe M, Jimenez-Garcia R. Gender Differences in the Prevalence and Characteristics of Pain in Spain: Report from a Population-Based Study. Pain Med. 2019 Dec 1;20(12):2349-2359. doi: 10.1093/pm/pnz004. PMID 30789640
- [Result] Fierro A, Perez-Roji G, Blanco A, Lopez P, Andres M, Gonzalez-Quintanilla V, Perez-Pereda S, Fontanillas N, Pascual J. Headache as main reason for consultation to a hospital Emergency Department in Spain: a prospective study. Neurologia (Engl Ed). 2021 May 31:S0213-4853(21)00089-X. doi: 10.1016/j.nrl.2021.03.015. Online ahead of print. English, Spanish. PMID 34083062
- [Result] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949